CLINICAL TRIAL: NCT00678964
Title: Multicentre Randomised Phase II Trial of Erlotinib Versus Carboplatin/Vinorelbine in Elderly Patients (=/> 70 Years) With Advanced Non-Small Cell Lung Cancer
Brief Title: Erlotinib Versus Carboplatin/Vinorelbine in Elderly Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Acronym: TIE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LungenClinic Grosshansdorf (Other)
Responsible Party: Dr. Martin Reck, Hospital Grosshansdorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2005-005827-32; ML19747
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Elderly patients
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Vinorelbine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Erlotinib
- B (Active Comparator)
  Interventions: Drug: Vinorelbine and Carboplatin

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150 mg, p.o., once daily
  Other Names: Tarceva
  Arms: A
Drug: Vinorelbine and Carboplatin — Vinorelbine 25 mg/m2, i.v., day 1 and 8 of every cycle (21 days) plus carboplatin AUC 5, i.v., day 1 of every cycle
  Other Names: Navelbine; Carboplat
  Arms: B

SUMMARY:
60% of all malignant diseases occur in patients who are 65 years or older. For these patients, aggressive treatments are often not suitable due to reduced life-expectancy, reduced general condition, comorbidities, and reduced vital functions which can lead to increased adverse effects of chemotherapy. Therefore, it is important to investigate alternative therapy options for elderly patients.

Erlotinib is an orally applied medication which is associated with reasonable toxicity. This targeted agent may prove an effective and well-tolerated first-line therapy in elderly patients with advanced non small cell lung cancer.

Therefore, the aim of this study is to investigate the progression-free survival of the combination of vinorelbine and carboplatin in comparison to erlotinib. Given that there will be no significant reduction of efficiency this may provide elderly patients of more than 70 years of age with an active oral substance without subjecting them to the sometimes severe adverse effect of the chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytological proven NSCLC, stage lll b (with pleural effusion) or stage lV.
* Tumour is locally advanced and not suitable for surgery and radiotherapy is not indicated.
* Neither cytostatic nor immunological pre-treatment
* Age >70 years
* At least one measurable lesion (RECIST criteria) that was not previously irradiated
* ECOG Performance Status 0-1
* Life expectancy > 3 month
* Adequate bone marrow function: ANC > 1.5 x 109/L, Platelets > 100 x 109/L
* Adequate liver function: Total Bilirubin < 1.5 x ULN, GOT/GPT< 3 x ULN (existent liver metastases < 5 x ULN)
* Adequate renal function:creatinine clearance > 45 ml/min (calculated according to Cockroft-Gault)
* Fertile men must agree to use an effective method of birth control while participating in this study
* Signed written informed consent

Exclusion Criteria:

* Uncontrolled metastasis in the CNS
* Acute, heavy uncontrolled infection
* Any other serious concomitant disease or medical condition, which could interfere with participating in this study
* Severe hypersensitivity to Erlotinib or any other component
* Hypersensitivity to Carboplatin and/or other platinum compounds
* Hypersensitivity to Vinorelbin or other Vinca-alkaloids
* Patients with a history of other active malignancy in the past 5 years (with the exception of carcinoma in situ of the cervix, non melanomatous skin cancers or local prostate carcinoma that was surgically treated successfully) are excluded.
* Participation in another clinical trial with any investigational drug at the same time or within 30 days prior to registration
* Psychological, familial, social or geographical situations limiting the compliance with the study requirements

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the progression free survival rate with the first-line therapy | Tumour assessment every other cycle (interval of 42 days)

SECONDARY OUTCOMES:
Duration of remission | Tumour assessment every other cycle (interval of 42 days)
1-year survival | 1 year
Overall survival | End of study
Response rate (CR/RR) | Tumour assessment every other cycle (interval of 42 days)
Quality of life, improvement of symptoms (FACT-L) | Every other cycle (interval of 42 days)
Simplified Charlsons´Comorbidity Score | baseline
Safety and Tolerability | continously

CONTACTS AND LOCATIONS:
Overall Officials: Martin Reck, Dr., Principal Investigator — LungenClinic Grosshansdorf
Locations (40):
- Germany (40):
  - Gemeinschaftspraxis, Augsburg
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Charité - Campus Benjamin Franklin, Berlin
  - Helios Klinikum Emil von Behring, Berlin
  - Evangelische Lungenklinik Berlin, Berlin
  - Evang. Krankenhaus Bielefeld, Bielefeld
  - Johanniter-Krankenhaus Bonn, Bonn
  - Gemeinschaftspraxis, Celle
  - Malteser Krankenhaus St. Hildegardis Köln, Cologne
  - Fachkrankenhaus Coswig, Coswig
  - Fachklinik Diekholzen, Diekholzen
  - Klinikum Donaustauf, Donaustauf
  - Katholisches Klinikum Duisburg, Duisburg
  - Marien Hospital Düsseldorf, Düsseldorf
  - Universitätsklinik Essen, Essen
  - Klinikum Essen-Mitte, Essen
  - Krankenhaus Nordwest GmbH, Frankfurt am Main
  - Asklepios Fachkliniken München-Gauting, Gauting
  - Schwerpunktpraxis Onkologie, Goslar
  - Georg-August-Universität Göttingen, Göttingen
  - Universitätsklinikum der Ernst-Moritz Arndt Universität Greifswald, Greifswald
  - Krankenhaus Großhansdorf, Großhansdorf
  - Allgemeines Krankenhaus Harburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Universitätsklinik des Saarlandes, Homburg/Saar
  - Klinikum der Friedrich-Schiller-Universität, Jena
  - Klinikum Kassel, Kassel
  - Klinikum Leverkusen gGmbH, Leverkusen
  - Klinik Löwenstein gGmbH, Löwenstein
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Katholisches Klinikum Mainz, Mainz
  - Klinikum der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Mannheim gGmbH, Mannheim
  - Zweckverband Kliniken im Mühlenkreis, Minden
  - Medizinische Klinik - Innenstadt, München
  - Ruppiner Kliniken GmbH, Neuruppin
  - Johanniter-Krankenhaus im Fläming gGmbH, Treuenbrietzen
  - Universitätsklinikum Ulm, Ulm